CLINICAL TRIAL: NCT07009951
Title: Acute Clinical Outcomes Following the Implementation of Virtual Reality (VR) in the Electrophysiology Laboratory
Brief Title: Impact of Virtual Reality in Cardiac Electrophysiology
Status: Recruiting | Type: Observational
Sponsor: University of Calabria (Other)
Responsible Party: Principal Investigator, Antonio Curcio, Professor, University of Calabria
Other Study IDs: 60/2025
Record Dates: First submitted 2025-05-15; First posted 2025-06-08 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Virtual reality Group: Patients who receive a virtual reality headset that provides an immersive environment, such as natural landscapes accompanied by relaxing music. The use of VR will begin at least five minutes before the start of the procedure to allow the patient to acclimate. The headset will remain in use throughout the entire procedure, unless complications arise (e.g., nausea or significant discomfort).
  Interventions: Device: Virtual reality
- Control Group (Standard Sedation): Patients who receive standard sedation (e.g. midazolam and/or fentanyl at the operator's discretion, according to hospital protocol), in accordance with comfort and analgesia guidelines for cardiac pacing procedures.

INTERVENTIONS:
Device: Virtual reality — VR headset provides an immersive environment, such as natural landscapes accompanied by relaxing music. The use of VR will begin at least five minutes before the start of the procedure to allow the patient to acclimate. The headset will remain in use throughout the entire procedure, unless complications arise (e.g., nausea or significant discomfort).
  Groups: Virtual reality Group

SUMMARY:
Pain during pacemaker or defibrillator implantation can increase patient discomfort, anxiety, and the need for deeper sedation. Using virtual reality (VR) as a non-pharmacological distraction tool may help reduce perceived pain, stabilize vital signs, and improve the overall patient experience. This prospective, single-center study evaluates whether adding VR to standard sedation lowers pain levels compared to sedation alone. Patients undergoing device implantation will be randomized to either group, with pain and vital signs monitored throughout the procedure. The study also explores patient satisfaction, adverse effects, and the potential of VR to support same-day discharge after minimally invasive procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patients who are candidates for pacemaker (PM) or implantable cardioverter-defibrillator (ICD) implantation, including new devices such as leadless PM and subcutaneous ICD (S-ICD).
* Ability to provide written informed consent.
* Ability to understand the use of the VR headset and express a pain score using the NRS scale.

Exclusion Criteria:

* Severe cognitive, psychiatric or neurological disorders that impair understanding or collaboration in the study.
* Visual and/or auditory and inner ear disorders or severe vertigo that could be aggravated by VR.
* Allergies or known adverse reactions to standard sedative therapies provided for in the protocol (e.g. midazolam) if essential for the procedure.
* Inability to correctly position the VR headset (e.g. severe facial deformities, recent trauma to the craniofacial area).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥18 years, eligible for implantation of cardiac pacing devices, able to provide informed consent and report their level of pain.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain and discomfort | during electrophysiology procedures
  To evaluate the difference in pain perception between a group using virtual reality (VR) and a control group subjected only to standard sedation, measured using the Numeric Rating Scale (NRS). The NRS is a self-reported scale ranging from 0 (no pain) to 10 (worst possible pain), where higher scores indicate greater pain and discomfort. The NRS will be recorded at the end of the procedure, referring to the pain experienced during the entire electrophysiology procedure.
Systolic Blood Pressure | during electrophysiology procedures
  To compare the change in systolic blood pressure (mmHg) during the procedure between the virtual reality (VR) group and the control group receiving standard sedation. Measurements will be taken at baseline, 15, 30, 45, and 60 minutes, and at the end of the procedure. The difference between groups will be assessed at each time point.
Heart Rate | during electrophysiology procedures
  To compare the change in heart rate (beats per minute) during the procedure between the virtual reality (VR) group and the control group receiving standard sedation. Measurements will be taken at baseline, 15, 30, 45, and 60 minutes, and at the end of the procedure. The difference between groups will be assessed at each time point.
Respiratory Rate | during electrophysiology procedures
  To compare the change in respiratory rate (breaths per minute) during the procedure between the virtual reality (VR) group and the control group receiving standard sedation. Measurements will be taken at baseline, 15, 30, 45, and 60 minutes, and at the end of the procedure. The difference between groups will be assessed at each time point.
Oxygen Saturation | during electrophysiology procedures
  To compare the change in oxygen saturation (SpO₂, %) during the procedure between the virtual reality (VR) group and the control group receiving standard sedation. Measurements will be taken at baseline, 15, 30, 45, and 60 minutes, and at the end of the procedure. The difference between groups will be assessed at each time point.

SECONDARY OUTCOMES:
Patient satisfaction | during electrophysiology procedures
  To evaluate patient satisfaction with the overall experience of the procedure. Satisfaction will be assessed using a structured questionnaire at the end of the procedure. Results will be expressed as a percentage score from 0% to 100%, where higher percentages indicate greater satisfaction. The satisfaction level will be categorized as follows:
  0-20%: Very unsatisfied 21-40%: Unsatisfied 41-60%: Neither satisfied nor unsatisfied 61-79%: Satisfied 80-100%: Very satisfied
Hospital stay length | through study completion, an average of 7 days
  To evaluate whether the use of virtual reality (VR) during electrophysiology procedures can contribute to a reduction in hospital stay, potentially allowing early discharge in some cases. The outcome will be measured as the mean number of days of hospital stay, and the difference between the VR group and the control group will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- "Annunziata" Hospital, Cosenza, Italy

IPD SHARING:
Plan to Share IPD: No